CLINICAL TRIAL: NCT00781625
Title: Probiotics/Lactobacillus as a Prophylactic Aid in Recurrent Bacterial Cystitis in Women. A Randomized, Prospective, Double-Blinded, Placebo Controlled, Multi-Center Study.
Brief Title: Probiotics as a Prophylactic Aid in Women With Recurrent Urinary Tract Infections (UTI's)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Akershus (Other)
Collaborators: St. Olavs Hospital (Other); Karolinska Institutet (Other); University of Oslo (Other); Folkehelsa (Unknown)
Responsible Party: MD Caroline Ursin Skagemo, Urologisk avdeling, Akershus Universitetssykehus HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S-08458d (REK); 08/7922(Shdir)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Urinary Tract Infections
Keywords: probiotics; QoL; inflammation; nutritional factors; prophylactic aid; Lactobacillus rhamnosus GR-1; Lactobacillus reuteri RC-14; Recurrent lower UTI in women
MeSH Terms: conditions — Urinary Tract Infections; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Probiotic vaginal capsules (Active Comparator): Probiotic vaginal capsule, placebo oral capsule
  Interventions: Dietary Supplement: UREX-cap-5
- placebo (Placebo Comparator): placebo oral capsule, placebo vaginal capsule
  Interventions: Dietary Supplement: Placebo Y cap G-3
- Probiotic oral capsules (Active Comparator): Probiotic oral capsules, placebo vaginal capsules
  Interventions: Dietary Supplement: UREX-cap-5

INTERVENTIONS:
Dietary Supplement: UREX-cap-5 — Size 3, white/white capsule, each containing 180 mg of a standardized, light beige fine powder consisting of freeze-dried cultures of: Lactobacillus rhamnosus, GR-1® (50%) Lactobacillus reuteri, RC-14® (50%) Ingredients Powder: Cultures, glucose anhydrate, potato starch, microcrystalline cellulose and magnesium stearate. Capsule: Gelatine, titanium dioxide Concentration Minimum of 5.4 billion (5.4 x 109) Colony Forming Units per capsule by end of bulk shelf life. Application For use as a dietary supplement. Packaging 20,000 capsules packaged in heat-sealed foil pouch.
  Arms: Probiotic oral capsules
Dietary Supplement: UREX-cap-5 — Size 3, white/white capsule, each containing 180 mg of a standardized, light beige fine powder consisting of freeze-dried cultures of: Lactobacillus rhamnosus, GR-1® (50%) Lactobacillus reuteri, RC-14® (50%) Ingredients Powder: Cultures, glucose anhydrate, potato starch, microcrystalline cellulose and magnesium stearate. Capsule: Gelatine, titanium dioxide Concentration Minimum of 5.4 billion (5.4 x 109) Colony Forming Units per capsule by end of bulk shelf life. Application For use as a dietary supplement. Packaging 20,000 capsules packaged in heat-sealed foil pouch.
  Arms: Probiotic vaginal capsules
Dietary Supplement: Placebo Y cap G-3 — Size 3, white/white capsule, each contaiing180 mg placebo blended powder. Daily oral and vaginal intake for a total duration of 6 months
  Arms: placebo

SUMMARY:
To investigate if administration of probiotics, either orally or vaginally,

* Can reduce the number of episodes of acute bacterial cystitis and/or
* Has tolerable adverse effect profile
* Improves general QoL in these women
* Improves the immune function and other physiological stress markers
* Reduces inflammation in urinary bladder epithelium

DETAILED DESCRIPTION:
Chronic recurrent bacterial cystitis is a condition that is disabling to a great extent and which influences quality of life and freedom of movement. The episodes can be painful, and lead to extensive use of antibiotics, which in itself promotes development of bacterial strains increasingly resistant to antibiotics, but do not prevent relapses. Almost all cystitis' in women are ascending infections from bacteria in the vagina, following colonization from the rectum. There have, however, been reported indications that there may be bacteria colonies within the urothelium that might give rise to relapses of the infections, rather than pure reinfection from ascending pathogens.

Probiotics are cultures of viable microorganisms, which show a positive effect on the general condition of the host when administered. Among the lactic acid bacteria (LAB), lactobacilli are the most commonly used for probiotics, and they have an excellent safety record. In terms of UTI, weekly or twice weekly intravaginal instillation of Lactobacillus strains GR-1 and B-54 have led to reduced recurrences. This concept has been supported by a 2006 pilot study showing that intravaginal administration of Lactobacillus crispatus GAI 98322 every two days for one year, had the potential to reduce the UTI recurrences. Another approach has been taken whereby lactobacilli are administered orally with a view of simulating how the pathogens reach the vagina. The studies have shown that L. rhamnosus GR-1 and L. reuteri (formerly fermentum) RC-14 can reach the vagina after daily oral ingestion, and they can lower the bacterial and yeast pathogen numbers.

The aim of the study is to try to normalize the vaginal bacteriological milieu so that the more pathogenic subpopulation of bacteria strains are displaced and are less likely to cause UTI.

ELIGIBILITY:
Inclusion Criteria:

* women 18-70 years old
* spontaneous urination
* > 3 UTI's previous year
* no ongoing prophylactic antibiotic treatment

Exclusion Criteria:

* > 50 ml residual urine
* neurological bladder disease
* known neoplasia, kidney stone or urinary tract abnormalities
* use og indwelling catheter
* pregnancy
* diabetes
* infrequent voiding pattern
* symptoms that indicate interstitial cystitis
* creatinin > 250 micmol/L
* participating in other clinical trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in number og episodes og lower UTI | 6 months intervention period
Improvement of QOL | 6 months intervention period

SECONDARY OUTCOMES:
Improvement of immune function | 6 months
Effects are non-dependant og nutritional status | 6 month2
Effects are non-dependant of known factors contributing til UTI's | 6 months
Decreases inflammation in the urinary bladder epithelium | 6 months
Normalizes vaginal microflora | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline U Skagemo, MD, Principal Investigator — Akershus Universitetssykehus HF; Gunn Iren Meling, PhD. MD, Study Director — Akershus Universitetssykehus HF
Locations (2):
- Norway (2):
  - Akershus Universitetssykehus HF, Lørenskog, Akershus
  - St.Olavs Hospital, Trondheim